CLINICAL TRIAL: NCT01088399
Title: The Global Hypopituitary Control and Complications Study
Brief Title: A Prospective Observational Study of Effect of Somatropin on Growth Hormone Deficient Adults
Acronym: HypoCCS
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 6448; B9R-MC-GDGA (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-02-25; First posted 2010-03-17 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Hypopituitarism; Pituitary Insufficiency; Growth Hormone Deficiency, Adult
MeSH Terms: conditions — Hypopituitarism; Dwarfism, Pituitary | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA Addendum - implemented in Germany only. Germany: DNA sample is kept, if participant consented to German DNA Addendum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Somatropin replacement treatment: Adult participants with growth hormone deficiency receiving somatropin replacement treatment.
  Interventions: Drug: Somatropin (rDNA origin)
- No treatment: Adult participants with growth hormone deficiency receiving no somatropin replacement treatment.

INTERVENTIONS:
Drug: Somatropin (rDNA origin) — Dose, frequency and duration are at discretion of attending physician, and determined on an individual basis.
  Other Names: Humatrope; LY137998
  Groups: Somatropin replacement treatment

SUMMARY:
The Hypopituitary Control and Complications Study "HypoCCS" is a prospective, open label, global, multicentre, observational study on routine clinical care of adults with growth hormone deficiency occurring either isolated or in combination with other pituitary hormone deficiencies. The objective of this observational study is to evaluate long-term safety and health outcomes for adult growth hormone deficient participants with or without somatropin replacement therapy. As an observational study, data are collected only as provided at the discretion of the attending physician. The participant enrolled meet the criteria of growth hormone deficiency in adults as per the Humatrope label in the country where their attending physician practices, and this diagnosis is at the discretion of the attending physician. The decision to receive somatropin or remain untreated is made by the participant in consultation with their attending physician.

While treatment of adult growth hormone deficient participants with somatropin has been shown to be safe and effective in clinical trials of 18 months duration, this observational study aims to provide information on health outcome and replacement therapy over longer periods of time for a larger number of participants in the context of the overall disease environment.

ELIGIBILITY:
Inclusion Criteria:

- Adult growth hormone deficiency as per the local Humatrope label and as judged by the attending physician

Exclusion Criteria:

- As per the local Humatrope label and as judged by the attending physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinics, private practices
Sampling Method: Non-Probability Sample
Enrollment: 10673 (Actual)
Dates: Start 2002-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company

REFERENCES:
- [Derived] Mo D, Blum WF, Rosilio M, Webb SM, Qi R, Strasburger CJ. Ten-year change in quality of life in adults on growth hormone replacement for growth hormone deficiency: an analysis of the hypopituitary control and complications study. J Clin Endocrinol Metab. 2014 Dec;99(12):4581-8. doi: 10.1210/jc.2014-2892. PMID 25233155
- [Derived] Mo D, Hardin DS, Erfurth EM, Melmed S. Adult mortality or morbidity is not increased in childhood-onset growth hormone deficient patients who received pediatric GH treatment: an analysis of the Hypopituitary Control and Complications Study (HypoCCS). Pituitary. 2014 Oct;17(5):477-85. doi: 10.1007/s11102-013-0529-6. PMID 24122237
- [Derived] Shimatsu A, Tai S, Imori M, Ihara K, Taketsuna M, Funai J, Tanaka T, Teramoto A, Irie M, Chihara K. Efficacy and safety of growth hormone replacement therapy in Japanese adults with growth hormone deficiency: a post-marketing observational study. Endocr J. 2013;60(10):1131-44. doi: 10.1507/endocrj.ej13-0083. Epub 2013 Jul 4. PMID 23823978
- [Derived] Attanasio AF, Jung H, Mo D, Chanson P, Bouillon R, Ho KK, Lamberts SW, Clemmons DR; HypoCCS International Advisory Board. Prevalence and incidence of diabetes mellitus in adult patients on growth hormone replacement for growth hormone deficiency: a surveillance database analysis. J Clin Endocrinol Metab. 2011 Jul;96(7):2255-61. doi: 10.1210/jc.2011-0448. Epub 2011 May 4. PMID 21543424

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were initially enrolled in 2 regional observational studies (B9R-EW-GDDQ [GDDQ] initiated in 1997 and B9R-MC-GDEE [GDEE] in 1998) which were merged into the global Study B9R-MC-GDGA (GDGA, NCT01088399) in 2002. This record spans approximately 15 years from the initial enrollment in regional studies to completion of Study GDGA.
Groups:
- Somatropin Treated: Participants received somatropin therapy dosed according to the local product label during the study. No form of intervention was imposed on the participants.
- Untreated: Participants did not receive somatropin therapy during the study. No form of intervention was imposed on the participants.
- FG002: It is not known whether participants did or did not receive somatropin therapy during the study. No form of intervention was imposed on the participants.
Period: Overall Study
Arm/Group | Somatropin Treated | Untreated | FG002
Started | 8716 | 1655 | 302
Completed | 1595 | 308 | 21
Not Completed | 7121 | 1347 | 281
Not completed — Adverse Event | 211 | 16 | 0
Not completed — Death | 204 | 45 | 0
Not completed — Lack of Efficacy | 298 | 7 | 5
Not completed — Lost to Follow-up | 1070 | 278 | 58
Not completed — Physician Decision | 531 | 88 | 16
Not completed — Withdrawal by Subject | 544 | 195 | 33
Not completed — Change to or start of somatropin therapy | 234 | 17 | 12
Not completed — Sponsor decision | 1573 | 298 | 7
Not completed — Protocol Violation | 10 | 1 | 0
Not completed — Enrollment criteria not met | 48 | 119 | 70
Not completed — Study summary visit not completed | 2398 | 283 | 80

BASELINE CHARACTERISTICS:
Groups:
- Unknown: It is unknown whether participants did or did not receive somatropin therapy during the study. No form of intervention was imposed on the participants.
- Total: Total of all reporting groups
Arm/Group | Somatropin Treated | Untreated | Unknown | Total
Number analyzed (Participants) | 8716 | 1655 | 302 | 10673
Age, Customized [Number; unit: participants]
  <20 years | 421 | 36 | 10 | 467
  20 years to <30 years | 1258 | 152 | 36 | 1446
  30 years to <40 years | 1475 | 173 | 54 | 1702
  40 years to <50 years | 1975 | 318 | 76 | 2369
  50 years to <60 years | 2048 | 379 | 74 | 2501
  60 years to <70 years | 1116 | 324 | 38 | 1478
  >=70 years | 421 | 272 | 13 | 706
  unknown | 2 | 1 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4158 | 714 | 155 | 5027
  Male | 4558 | 941 | 147 | 5646
Race/Ethnicity, Customized [Number; unit: participants]
  African Descent | 226 | 96 | 14 | 336
  Caucasian | 6058 | 1080 | 236 | 7374
  East/Southeast Asian | 460 | 129 | 7 | 596
  Hispanic | 153 | 55 | 16 | 224
  Western Asian | 24 | 5 | 3 | 32
  Other | 38 | 10 | 2 | 50
  Declined To Provide | 387 | 82 | 12 | 481
  Unknown | 1370 | 198 | 12 | 1580
Region of Enrollment [Number; unit: participants]
  Austria | 77 | 1 | 1 | 79
  Belgium | 55 | 1 | 0 | 56
  Canada | 63 | 51 | 0 | 114
  Czech Republic | 77 | 5 | 0 | 82
  Denmark | 151 | 5 | 0 | 156
  France | 452 | 218 | 6 | 676
  Germany | 553 | 87 | 19 | 659
  Hungary | 102 | 2 | 0 | 104
  Iceland | 10 | 1 | 1 | 12
  Italy | 1242 | 64 | 49 | 1355
  Japan | 407 | 102 | 0 | 509
  Norway | 17 | 0 | 0 | 17
  Spain | 427 | 55 | 2 | 484
  Sweden | 355 | 3 | 2 | 360
  Netherlands | 460 | 1 | 0 | 461
  United Kingdom | 538 | 15 | 6 | 559
  United States | 3730 | 1044 | 216 | 4990
Growth Hormone Deficiency (GHD) Onset Type [Number; unit: participants]
  Adult | 6968 | 1422 | 247 | 8637
  Childhood | 1702 | 194 | 29 | 1925
  Unknown | 46 | 39 | 26 | 111
Insulin-like Growth Factor-I (IGF-I) [Mean (Standard Deviation); unit: micrograms per liter (mcg/L)] — Participants with available IGF-I data at baseline (n=5531, 1009, 194 with 6734 total participants). IGF-I is primary mediator of growth hormone (GH) and is used to monitor GH effectiveness, treatment adherence and IGF-I excess.
  micrograms per liter (mcg/L) | 100.4 (78.0) | 75.0 (55.3) | 95.5 (63.7) | 96.4 (75.2)
IGF-I Standard Deviations Score (SDS) [Mean (Standard Deviation); unit: standard deviation scores] — Participants with available IGF-I SDS data at baseline (n=3743, 645, 113 with 4501 total participants). IGF-I is primary mediator of growth hormone (GH) and is used to monitor GH effectiveness, treatment adherence and IGF-I excess. As endogenous levels of GH, thereby IGF-I, decline throughout adulthood values are converted to age and gender adjusted standard deviation scores (SDS) based on general population normal data. The SDS is the number of standard deviations a subjects IGF-I concentration is different from the general population mean, either positive or negative.
  standard deviation scores | -2.72 (2.23) | -2.82 (1.97) | -2.39 (2.03) | -2.73 (2.19)
Maximum Growth Hormone (GH) Peak on Stimulation Test [Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)] — Participants with available maximum GH peak data at baseline (N=1175, 103, 51 with 1329 total participants analyzed). Maximum GH peak levels in response to medication (such as insulin or growth hormone releasing hormone (GHRH) plus arginine) or other intervention (such as exercise) was used to measure the ability of the pituitary gland to release GH and to diagnose and determine severity of GH deficiency. Severe GH deficiency in adults is a peak GH response of <3 milligrams/liter in response to an insulin tolerance test and is an accepted criterion for GH replacement therapy in adults.
  nanograms per milliliter (ng/mL)
    GHRH + Arginine (Arg, n=1175, 103, 51, 1329) | 2.5 (3.5) | 5.2 (8.1) | 4.4 (8.1) | 2.8 (4.4)
    Any test except GHRH + Arg (n=6579;1178;168;7925) | 1.1 (1.9) | 2.0 (3.7) | 5.2 (6.7) | 1.3 (2.5)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Participants with available BMI data at baseline (n=8263, 1452, 268, with 9983 total participants). Body mass index (BMI) is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 29.7 (7.0) | 29.9 (7.0) | 30.0 (6.9) | 29.7 (7.0)
Diagnosis Leading to GHD [Number; unit: participants] — Participants with available diagnosis designation at baseline (n=8670, 1616, 276, with 10562 total participants). Other less common specified diagnoses contains participants who had histories including cranial irradiation, empty sella, hypophysitis, congenital defect resulting in GHD.
  participants
    Pituitary adenoma | 3769 | 865 | 79 | 4713
    Craniopharyngioma | 973 | 125 | 24 | 1122
    Other Tumor | 653 | 137 | 7 | 797
    Idiopathic | 1381 | 177 | 88 | 1646
    Pituitary hemorrhage/brain injury | 455 | 59 | 4 | 518
    Other less common specified diagnoses | 1027 | 198 | 79 | 1304
    Causes other than listed above | 458 | 94 | 21 | 573

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant Adverse Events
Description: A summary of all reported serious adverse events (SAE) and other adverse events regardless of causality are provided in the Adverse Events module of this record.
Time Frame: Baseline to study completion (approximately 10 years)
Population: All participants with baseline and at least 1 post-baseline visit whose study therapy was known (treated or untreated).
Measure: Number; unit: percentage of participants
Arm/Group | Somatropin Treated | Untreated
Number analyzed (Participants) | 8420 | 1269
percentage of participants
  Death | 2.58 | 3.78
  Malignancy | 4.0 | 5.3
  Myocardial Infarction | 0.8 | 1.4

2. Secondary Outcome: Cardiovascular Risk Factor-Change From Baseline in Body Mass Index (BMI)
Description: Change in BMI was used as an indicator of cardiovascular risk. Body mass index (BMI) is an estimate of body fat based on body weight divided by height squared.
Time Frame: Baseline, interim time point (5 years), and study completion (10 years)
Population: All participants with baseline and at least 1 post-baseline visit whose study therapy was known (treated or untreated) and had BMI data.
Measure: Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)
Arm/Group | Somatropin Treated | Untreated
Number analyzed (Participants) | 8263 | 1452
kilogram per square meter (kg/m^2)
  Change in BMI at 5 years (n=2541, 218) | 0.63 (3.15) | -0.10 (3.25)
  Change in BMI at 10 years (n=884, 64) | 1.14 (3.67) | -0.32 (2.67)

3. Secondary Outcome: Cardiovascular Risk Factor-Change From Baseline in Systolic (SBP) and Diastolic Blood Pressure (DBP)
Description: Change in SBP and DBP were used as an indicator of cardiovascular risk.
Time Frame: Baseline, interim time point (5 years), and study completion (10 years)
Population: All participants with baseline and at least 1 post-baseline visit whose study therapy was known (treated or untreated) and BP data.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Somatropin Treated | Untreated
Number analyzed (Participants) | 8258 | 1546
millimeters of mercury (mmHg)
  Change in SBP at 5 years (n=2746, 272) | 1.04 (17.49) | -0.48 (18.88)
  Change in SBP at 10 years (n=960, 73) | 1.98 (18.81) | 3.71 (20.04)
  Change in DBP at 5 years (n=2740, 272) | -0.85 (11.11) | -0.76 (11.71)
  Change in DBP at 10 years (n=955, 73) | -1.23 (11.85) | -2.84 (13.37)

4. Secondary Outcome: Cardiovascular Risk Factor-Change From Baseline in Cholesterol and Triglycerides
Description: Change from baseline in total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C) and triglycerides were used as an indicator of cardiovascular risk and are presented.
Time Frame: Baseline, interim time point (5 years), and study completion (10 years)
Population: All participants with baseline and at least 1 post-baseline visit whose study therapy was known (treated or untreated) and had cholesterol or triglyceride data.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Somatropin Treated | Untreated
Number analyzed (Participants) | 6327 | 1171
milligrams per deciliter (mg/dL)
  Change in TC at 5 years (n=1865, 184) | -13.0 (45.74) | -14.6 (46.02)
  Change in TC at 10 years (n=668, 56) | -17.9 (52.87) | -43.1 (55.81)
  Change in HDL-C at 5 years (n=1667, 176) | 1.47 (16.67) | -0.54 (13.82)
  Change in HDL-C at 10 years (n=615, 51) | 5.00 (17.40) | 0.39 (14.70)
  Change in LDL-C at 5 years (1435, 166) | -10.7 (41.32) | -11.5 (35.91)
  Change in LDL-C at 10 years (n=522, 47) | -16.4 (44.05) | -29.3 (41.44)
  Change in Triglycerides at 5 years (n=1581, 178) | -9.51 (99.67) | -0.85 (115.7)
  Change in Triglycerides at 10 years (n=571, 51) | -16.4 (107.8) | -55.8 (90.12)

5. Secondary Outcome: Cardiovascular Risk Factor-Change From Baseline in Waist Circumference
Description: Change in waist circumference was used as an indicator of cardiovascular risk.
Time Frame: Baseline, interim time point (5 years), and study completion (10 years)
Population: All participants with baseline and at least 1 post-baseline visit whose study therapy was known (treated or untreated) and had waste circumference data.
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Somatropin Treated | Untreated
Number analyzed (Participants) | 6263 | 1005
centimeters (cm)
  Change in circumference at 5 years (n=1719, 133) | 0.85 (9.06) | 0.10 (8.52)
  Change in circumference at 10 years (n=610, 34) | 3.57 (10.22) | 3.03 (7.76)

6. Secondary Outcome: Percentage of Participants Experiencing a Bone Fracture (Fracture Incidence)
Time Frame: Baseline through 10 years
Population: All participants with baseline and at least 1 post-baseline visit and who provided bone fracture information.
Measure: Number; unit: percentage of participants
Arm/Group | Somatropin Treated | Untreated | Unknown
Number analyzed (Participants) | 8420 | 1269 | 4
percentage of participants | 3.75 | 4.02 | 0.00

7. Secondary Outcome: Change From Baseline in the Total Z Score of the Disease-specific Module of the Questions of Life Satisfaction (QLS-H).
Description: QLS-H is a self-administered, weighted, quality of life (QoL) questionnaire consisting of 9 items developed for participants with growth hormone deficiency. Scores were corrected for age, gender, and country differences, and expressed as Z-scores based on country-specific reference ranges. Participants indicate how important a certain dimension of QoL is to them and are then questioned as to their degree of satisfaction with that dimension. Each item is rated on a 5-point Likert scale ranging from not important (1) to extremely important (5) and from dissatisfied (1) to very satisfied (5). The weighted score for the degree of satisfaction (weighted satisfaction) with a particular dimension=(importance - 1)x(2 x satisfaction - 5). Total Z-score is obtained by adding the individual item scores of the 9 dimensions, and range from -108 (representing very low satisfaction) to +180 (representing very high satisfaction).
Time Frame: Baseline, interim time point (5 years), and study completion (10 years)
Population: All participants with baseline and at least 1 post-baseline visit whose study therapy was known (treated or untreated) and has a Total Z Score.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Somatropin Treated | Untreated
Number analyzed (Participants) | 2142 | 332
Z-score
  Change in Total Z score at 5 years (n=475, 39) | 0.70 (1.46) | 0.21 (1.14)
  Change in Total Z score at 10 years (n=103, 3) | 0.53 (1.39) | -1.01 (1.49)

8. Other Pre Specified Outcome: Number of Participants Who Died While in the Study
Time Frame: Study enrollment up to approximately 10 years
Population: All participants with baseline and at least 1 post-baseline visit.
Measure: Number; unit: participants
Arm/Group | Somatropin Treated | Untreated | Unknown
Number analyzed (Participants) | 8420 | 1269 | 4
participants | 229 | 50 | 0

ADVERSE EVENTS:
Time Frame: Study enrollment up to approximately 10 years.
Description: All participants with baseline and at least 1 post-baseline visit.
Groups:
- EG002: It is unknown whether participants did or did not receive somatropin therapy during the study. No form of intervention was imposed on the participants.
Arm/Group | Somatropin Treated | Untreated | EG002
Serious Adverse Events (participants affected / at risk) | 1602/8420 | 288/1269 | 0/4
Other Adverse Events (participants affected / at risk) | 4912/8420 | 591/1269 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Somatropin Treated (N=8420) | Untreated (N=1269) | EG002 (N=4)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 5 (5) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 6 (6) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 13 (13) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 16 (17) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 7 (7) | 2 (2) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 6 (6) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 26 (28) | 11 (13) | 0 (0)
Atrial flutter (Cardiac disorders) | 4 (4) | 3 (3) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrioventricular dissociation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 5 (5) | 4 (4) | 0 (0)
Bundle branch block left (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 13 (13) | 3 (3) | 0 (0)
Cardiac failure (Cardiac disorders) | 13 (15) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 19 (22) | 10 (11) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 4 (4) | 0 (0)
Cardiomegaly (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 22 (23) | 7 (7) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 39 (41) | 12 (13) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 5 (5) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 6 (7) | 2 (2) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Subendocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 6 (6) | 1 (1) | 0 (0)
Wolff-parkinson-white syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arnold-chiari malformation (Congenital, familial and genetic disorders) | 2 (3) | 0 (0) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Diencephalic syndrome of infancy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmorphism (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Gene mutation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Porphyria (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 1 (2) | 1 (1) | 0 (0)
Endolymphatic hydrops (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 5 (5) | 2 (2) | 0 (0)
Addison's disease (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Adrenal disorder (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 29 (29) | 4 (4) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 54 (62) | 6 (7) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Carcinoid syndrome (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0)
Hyperadrenocorticism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperprolactinaemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Hypothalamo-pituitary disorder (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Lymphocytic hypophysitis (Endocrine disorders) | 5 (7) | 0 (0) | 0 (0)
Nelson's syndrome (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Pituitary cyst (Endocrine disorders) | 4 (4) | 0 (0) | 0 (0)
Pituitary enlargement (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Pituitary haemorrhage (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0)
Pituitary-dependent cushing's syndrome (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 11 (12) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Blindness unilateral (Eye disorders) | 1 (3) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 4 (4) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Scotoma (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 21 (22) | 3 (3) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Appendix disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic enteropathy (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 29 (30) | 7 (7) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 6 (6) | 2 (2) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 (13) | 4 (4) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 6 (7) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mesenteric occlusion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 33 (35) | 4 (4) | 0 (0)
Oesophageal dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 7 (9) | 4 (4) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peritoneal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary gland mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 7 (8) | 2 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 38 (45) | 4 (4) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 11 (13) | 4 (4) | 0 (0)
Chest discomfort (General disorders) | 5 (5) | 1 (1) | 0 (0)
Chest pain (General disorders) | 37 (41) | 9 (9) | 0 (0)
Chills (General disorders) | 1 (1) | 2 (2) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 48 (48) | 15 (15) | 0 (0)
Device failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 1 (2) | 0 (0)
Drug intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 0 (0)
Fibrosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (2) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic cyst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Hernia obstructive (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperpyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 2 (3) | 0 (0)
Implant site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Medical device pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ disorder (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 10 (14) | 3 (3) | 0 (0)
Oedema (General disorders) | 2 (2) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 3 (3) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0) | 0 (0)
Polyp (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pseudocyst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 27 (28) | 7 (8) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 3 (3) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 8 (8) | 3 (3) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 4 (4) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 21 (21) | 4 (4) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 2 (3) | 2 (2) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 2 (2) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 2 (2) | 0 (0)
Sarcoidosis (Immune system disorders) | 5 (7) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 12 (12) | 5 (5) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atypical mycobacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 11 (11) | 6 (7) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 19 (27) | 4 (5) | 0 (0)
Chronic sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Colostomy infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Corneal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Creutzfeldt-jakob disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Cystitis klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus hepatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 16 (19) | 3 (4) | 0 (0)
Echinococciasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Encephalitic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Encephalitis viral (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 5 (5) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Extradural abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gallbladder empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 43 (45) | 5 (8) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 13 (14) | 3 (5) | 0 (0)
Gastrointestinal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Incision site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 5 (5) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infectious peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 15 (15) | 5 (5) | 0 (0)
Infusion site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 5 (9) | 2 (2) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Meningitis (Infections and infestations) | 7 (7) | 3 (3) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Meningitis bacterial (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 6 (7) | 0 (0) | 0 (0)
Meningoencephalitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mycobacterium avium complex infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 3 (4) | 2 (2) | 0 (0)
Pelvic abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 95 (107) | 23 (28) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia herpes viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Post procedural pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Purulent discharge (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 26 (26) | 8 (8) | 0 (0)
Septic shock (Infections and infestations) | 7 (7) | 5 (5) | 0 (0)
Shunt infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 9 (9) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Subacute endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 22 (26) | 7 (8) | 0 (0)
Urosepsis (Infections and infestations) | 9 (11) | 2 (3) | 0 (0)
Viraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 16 (16) | 4 (4) | 0 (0)
Viral pericarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 7 (7) | 2 (2) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Delayed effects of radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 28 (28) | 5 (5) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 (6) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 7 (8) | 3 (3) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Graft complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 8 (8) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 4 (5) | 0 (0) | 0 (0)
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 8 (8) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 6 (7) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Meningitis chemical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Mountain sickness acute (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Open wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 9 (9) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Poisoning deliberate (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative adhesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 15 (15) | 2 (2) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 6 (6) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic lung injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 0 (0)
Uterine rupture (Injury, poisoning and procedural complications) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 0 (0)
Amniotic fluid volume increased (Investigations) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Anticoagulation drug level below therapeutic (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspiration bone marrow (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspiration pleural cavity (Investigations) | 1 (2) | 0 (0) | 0 (0)
Band neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood cortisol decreased (Investigations) | 4 (4) | 0 (0) | 0 (0)
Blood cortisol increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood electrolytes abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Bone density decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Bronchoscopy (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cardiac enzymes increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cortisol free urine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Drug level below therapeutic (Investigations) | 1 (1) | 0 (0) | 0 (0)
Drug level increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram change (Investigations) | 0 (0) | 1 (1) | 0 (0)
Endoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haematocrit increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 1 (1) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hysteroscopy (Investigations) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Immunosuppressant drug level decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1/4394 (1) | 0/745 (0) | 0/2 (0)
Smear cervix abnormal (Investigations) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Ureteroscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 44 (48) | 16 (18) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 15 (15) | 2 (2) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (9) | 0 (0) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 5 (6) | 3 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 13 (17) | 4 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (12) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 35 (44) | 11 (12) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 8 (9) | 1 (1) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1) | 0 (0)
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hip deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 20 (21) | 2 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 20 (25) | 5 (5) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
B-cell lymphoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (22) | 4 (5) | 0 (0)
Benign neoplasm of testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/4394 (1) | 0/745 (0) | 0/2 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Benign respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 (16) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Carotid body tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cns germinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 3 (3) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 0 (0) | 0 (0)
Craniopharyngioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dermatofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Endometrial cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Ewing's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Germ cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1) | 0 (0)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm of islets of langerhans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Mantle cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Medulloblastoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 (23) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (5) | 0 (0) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Mixed oligo-astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/4394 (1) | 0/745 (0) | 0/2 (0)
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 1 (1) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0)
Non-hodgkin's lymphoma stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Non-secretory adenoma of pituitary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Optic nerve neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/4025 (2) | 0/524 (0) | 0/2 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/4394 (0) | 1/745 (1) | 0/2 (0)
Pharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 3 (3) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 (24) | 8 (9) | 0 (0)
Pituitary tumour recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 115 (128) | 19 (19) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (5) | 0 (0) | 0 (0)
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 33/4394 (36) | 10/745 (10) | 0/2 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/4394 (1) | 0/745 (0) | 0/2 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/4394 (1) | 0/745 (0) | 0/2 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Secretory adenoma of pituitary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/4025 (2) | 0/524 (0) | 0/2 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/4025 (3) | 0/524 (0) | 0/2 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Balance disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Basilar artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid aneurysm rupture (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 7 (7) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 7 (7) | 0 (0) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cerebral cyst (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Cerebral disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 9 (9) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 15 (17) | 3 (3) | 0 (0)
Cerebral thrombosis (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 63 (73) | 16 (16) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 5 (5) | 1 (1) | 0 (0)
Coma hepatic (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 22 (25) | 8 (8) | 0 (0)
Dementia (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 13 (14) | 5 (5) | 0 (0)
Dysarthria (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 12 (13) | 2 (2) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 8 (8) | 0 (0) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 5 (5) | 3 (3) | 0 (0)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 22 (26) | 2 (3) | 0 (0)
Hemianopia (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Hemianopia heteronymous (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 9 (9) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 5 (5) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 5 (5) | 3 (3) | 0 (0)
Ivth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 5 (5) | 3 (3) | 0 (0)
Loss of consciousness (Nervous system disorders) | 5 (5) | 2 (3) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Mononeuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Moyamoya disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 4 (4) | 2 (2) | 0 (0)
Quadriplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Spinal cord oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 5 (5) | 1 (1) | 0 (0)
Subdural hygroma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 33 (36) | 16 (16) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 30 (34) | 4 (4) | 0 (0)
Tremor (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Viith nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Visual field defect (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Visual pathway disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Vith nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abnormal labour (Pregnancy, puerperium and perinatal conditions) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2/4025 (2) | 0/524 (0) | 0/2 (0)
Delivery (Pregnancy, puerperium and perinatal conditions) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 7/4025 (7) | 0/524 (0) | 0/2 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 2/4025 (2) | 0/524 (0) | 0/2 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (6) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 8 (8) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 14 (16) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 17 (18) | 3 (5) | 0 (0)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Drug dependence (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Drug dependence, postpartum (Psychiatric disorders) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 2 (4) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 13 (13) | 7 (7) | 0 (0)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Substance abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 6 (6) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 8 (9) | 0 (0) | 0 (0)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Crush syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 5 (5) | 0 (0) | 0 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydroureter (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 9 (10) | 2 (2) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 2 (3) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 12 (13) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 10 (11) | 6 (9) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 5 (5) | 2 (2) | 0 (0)
Renal mass (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 5 (5) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vesical fistula (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Adnexa uteri cyst (Reproductive system and breast disorders) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Adnexa uteri mass (Reproductive system and breast disorders) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Artificial menopause (Reproductive system and breast disorders) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 8/4394 (8) | 2/745 (2) | 0/2 (0)
Breast enlargement (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 2/4025 (2) | 0/524 (0) | 0/2 (0)
Endometrial disorder (Reproductive system and breast disorders) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Endometriosis (Reproductive system and breast disorders) | 2/4025 (2) | 0/524 (0) | 0/2 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1/4394 (1) | 0/745 (0) | 0/2 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Menopausal disorder (Reproductive system and breast disorders) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Menorrhagia (Reproductive system and breast disorders) | 2/4025 (2) | 0/524 (0) | 0/2 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Ovarian cyst (Reproductive system and breast disorders) | 8/4025 (9) | 1/524 (1) | 0/2 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Ovarian mass (Reproductive system and breast disorders) | 2/4025 (2) | 0/524 (0) | 0/2 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 1/4394 (2) | 0/745 (0) | 0/2 (0)
Prostatism (Reproductive system and breast disorders) | 1/4394 (1) | 0/745 (0) | 0/2 (0)
Prostatitis (Reproductive system and breast disorders) | 2/4394 (2) | 0/745 (0) | 0/2 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1/4394 (1) | 0/745 (0) | 0/2 (0)
Rectocele (Reproductive system and breast disorders) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Testicular atrophy (Reproductive system and breast disorders) | 1/4394 (1) | 0/745 (0) | 0/2 (0)
Uterine polyp (Reproductive system and breast disorders) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Uterine prolapse (Reproductive system and breast disorders) | 3/4025 (3) | 0/524 (0) | 0/2 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2/4025 (2) | 0/524 (0) | 0/2 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 3 (5) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Broncholithiasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 3 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 4 (4) | 0 (0)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 4 (4) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 3 (3) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (6) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 0 (0)
Alcohol use (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Abdominal panniculectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 2/4025 (2) | 0/524 (0) | 0/2 (0)
Adhesiolysis (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Adrenalectomy (Surgical and medical procedures) | 3 (3) | 0 (0) | 0 (0)
Aneurysm repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 7 (7) | 0 (0) | 0 (0)
Arterial bypass operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula operation (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0)
Bladder operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Brain operation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Breast lump removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Bunion operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cardiac ablation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Cardioversion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Carotid artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 5 (5) | 0 (0) | 0 (0)
Carpal tunnel decompression (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 8 (8) | 0 (0) | 0 (0)
Cholelithotomy (Surgical and medical procedures) | 3 (3) | 0 (0) | 0 (0)
Colectomy (Surgical and medical procedures) | 2 (2) | 1 (1) | 0 (0)
Colostomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 1 (1) | 1 (2) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 2 (2) | 1 (1) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Craniotomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Enterostomy closure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Ethmoid sinus surgery (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Explorative laparotomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Foot operation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Foraminotomy (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Gallbladder operation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Gastrectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 3 (3) | 1 (1) | 0 (0)
Haematoma evacuation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Haemodialysis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hernia hiatus repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
High frequency ablation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 11 (12) | 1 (2) | 0 (0)
Hip surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hypophysectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 6/4025 (6) | 0/524 (0) | 0/2 (0)
Ileostomy closure (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Implantable defibrillator insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Implantable defibrillator replacement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Incisional drainage (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Internal fixation of fracture (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc operation (Surgical and medical procedures) | 2 (3) | 0 (0) | 0 (0)
Intestinal resection (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 5 (6) | 1 (1) | 0 (0)
Knee operation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Lipoma excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Lithotripsy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Liver transplant (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Lung transplant (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Malignant breast lump removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Mastectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Mechanical ventilation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Medical device implantation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Meningeal repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Meningioma surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Meniscus operation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Meniscus removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Nasal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Open reduction of fracture (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Osteosynthesis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Ovarian cystectomy (Surgical and medical procedures) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Pancreatectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Parathyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Peripheral nerve decompression (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Pituitary gland radiotherapy (Surgical and medical procedures) | 5 (5) | 0 (0) | 0 (0)
Pituitary tumour removal (Surgical and medical procedures) | 19 (23) | 3 (3) | 0 (0)
Plastic surgery to the face (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Preoperative care (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Prostatic operation (Surgical and medical procedures) | 2/4394 (2) | 0/745 (0) | 0/2 (0)
Radiotherapy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Rectal prolapse repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Renal tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Salivary gland operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Shoulder arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Sigmoidectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Sinus antrostomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Sinus operation (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Skin graft (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Sphenoid sinus operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Spinal decompression (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 4 (4) | 0 (0) | 0 (0)
Spinal operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Splenectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Stent placement (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Subdural haematoma evacuation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 3 (3) | 0 (0) | 0 (0)
Thyroid operation (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 2 (2) | 1 (1) | 0 (0)
Toe operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Transfusion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 4/4394 (4) | 0/745 (0) | 0/2 (0)
Tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 3 (3) | 0 (0) | 0 (0)
Urethral repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Uterine dilation and curettage (Surgical and medical procedures) | 1/4025 (1) | 0/524 (0) | 0/2 (0)
Wound closure (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Wound treatment (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Aneurysm (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 5 (5) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Artery dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 21 (22) | 3 (3) | 0 (0)
Haematoma (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 7 (7) | 4 (5) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 19 (20) | 8 (10) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Infarction (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 5 (7) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 2 (4) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Vein disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Somatropin Treated (N=8420) | Untreated (N=1269) | EG002 (N=4)
Diarrhoea (Gastrointestinal disorders) | 165 (202) | 34 (41) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 167 (169) | 26 (26) | 0 (0)
Nausea (Gastrointestinal disorders) | 213 (242) | 24 (29) | 0 (0)
Asthenia (General disorders) | 206 (216) | 36 (42) | 0 (0)
Fatigue (General disorders) | 495 (524) | 75 (76) | 0 (0)
Oedema peripheral (General disorders) | 546 (624) | 27 (31) | 0 (0)
Influenza (Infections and infestations) | 198 (216) | 13 (14) | 0 (0)
Nasopharyngitis (Infections and infestations) | 176 (211) | 16 (16) | 0 (0)
Sinusitis (Infections and infestations) | 242 (322) | 22 (24) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 185 (234) | 28 (34) | 0 (0)
Weight increased (Investigations) | 185 (192) | 21 (21) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 194 (209) | 24 (24) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 263 (268) | 37 (37) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 144 (145) | 39 (39) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 742 (887) | 48 (54) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 347 (384) | 33 (35) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 236 (252) | 12 (12) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 184 (185) | 35 (35) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 164 (165) | 41 (41) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 276 (315) | 30 (38) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 181 (196) | 10 (11) | 0 (0)
Dizziness (Nervous system disorders) | 220 (238) | 40 (44) | 0 (0)
Headache (Nervous system disorders) | 533 (607) | 57 (66) | 0 (0)
Paraesthesia (Nervous system disorders) | 210 (233) | 4 (4) | 0 (0)
Depression (Psychiatric disorders) | 557 (590) | 54 (56) | 0 (0)
Insomnia (Psychiatric disorders) | 185 (192) | 22 (22) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 74/4394 (76) | 16/745 (16) | 0/2 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 182 (184) | 20 (20) | 0 (0)
Hypertension (Vascular disorders) | 630 (671) | 59 (61) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days